CLINICAL TRIAL: NCT05319028
Title: A Phase 2 Study of Mivavotinib in Biomarker-Defined Subgroups of Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Study of Mivavotinib (CB-659) in Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX-659-401
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Non-GCB/ABC Diffuse Large B-Cell Lymphoma; With and Without MyD88 and/or CD79B Mutations
Keywords: Mivavotinib; DLBCL; MyD88; CD79b; non-GCB; ABC; NHL; CB-659; Relapsed/Refractory
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Dosing Schedule (Experimental): Mivavotinib 100 mg once daily (QD)
  Interventions: Drug: Mivavotinib
- Induction Dosing Schedule (Experimental): Mivavotinib 120 mg QD for 14 days, then 80 mg QD starting Day 15
  Interventions: Drug: Mivavotinib

INTERVENTIONS:
Drug: Mivavotinib — oral tablet
  Other Names: CB-659

SUMMARY:
Study CX-659-401 is a multicenter, open-label, phase 2 study of mivavotinib to evaluate the single-agent activity of mivavotinib in patients with relapsed/refractory non-GCB/ABC DLBCL, incorporating ctDNA-based next-generation sequencing (NGS) to identify DLBCL patients harboring MyD88 and/or CD79B mutations within the study. This goal of this strategy is to evaluate its activity both in the cell-of-origin subgroup of non-GCB/ABC DLBCL and in the genetically defined subgroups of MyD88/CD79B-mutated and wild type DLBCL.

DETAILED DESCRIPTION:
Approximately 50 patients will be randomized 1:1 to one of two dose/schedule cohorts: one with a continuous dosing schedule (100 mg QD) and one with an induction dosing schedule (120 mg QD x 14 days, then 80 mg QD starting Day 15). Patients will receive treatment with mivavotinib until disease progression, unacceptable toxicity, withdrawal of consent, or death.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
3. Life expectancy of > 3 months
4. Histologically confirmed de novo or transformed non-GCB DLBCL.
5. Relapsed or refractory to ≥ 2 prior lines of chemotherapy based on standard of care
6. Patients should not have failed more than 5 prior lines of therapy
7. Must have [18F]Fluorodeoxyglucose-positron emission tomography (FDG-PET)-avid measurable disease that meets the size criteria per International Working Group (IWG) criteria.
8. Must have recovered from adverse events of prior anti-cancer therapy to severity ≤ Grade 1.
9. Adequate organ function as assessed by laboratory values.
10. If female of childbearing potential, agreement to use protocol specified contraception methods. If male, agreement to use an effective barrier method of contraception.

Exclusion Criteria:

1. DLBCL with central nervous system (CNS) involvement with active brain or leptomeningeal disease
2. Known human immunodeficiency (HIV; testing not required) or HIV-related malignancy
3. Known hepatitis B surface antigen positive or known or active hepatitis C infection
4. Prior autologous stem cell transplant (ASCT) or chimeric antigen receptor T-cell (CAR-T) cell infusion within 90 days of screening
5. Prior allogeneic stem cell transplantation
6. Unstable/inadequate cardiac function
7. Known gastrointestinal (GI) disease or GI procedure that interferes with swallowing/absorption of oral drug
8. Major surgery within 14 days before the first dose of study drug
9. Serious infection (bacterial/fungal/viral) requiring parenteral antibiotic/antiviral therapy for >5 days within 21 days prior to first dose of study drug
10. Treatment with high-dose corticosteroids for anticancer purposes within 7 days before the first dose of mivavotinib.
11. Use of medication known to be inhibitors or inducers of P-glycoprotein (P-gp) and/or Cytochrome P (CYP)3A
12. Female patients who are pregnant, lactating or breastfeeding.
13. Any radiation therapy within 3 weeks prior to first dose of study treatment.
14. Systemic anticancer treatment within 3 weeks before first dose of study treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as assessed by an independent radiology review committee (IRC) according to the 2014 International Working Group (IWG) Lugano Criteria (Cheson, 2014). | Start of treatment up to 21 months
  Overall response is defined as a complete response (CR) or partial response (PR). ORR is the proportion of participants who have overall responses.
Safety as measured by type, incidence, severity, seriousness, and study drug-relatedness of adverse events per Common Terminology Criteria for Adverse Events, version 5 | Start of treatment up to 21 months
  Type, incidence, severity, seriousness, and study drug-relatedness of AEs assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Duration of Response (DOR) Rate as assessed by an IRC according to the 2014 International Working Group (IWG) Lugano Criteria (Cheson, 2014). | Start of treatment up to 21 months
  DOR per IRC. DOR will be calculated as the time between the first documentation of partial response (PR) or a complete response (CR) to the first documentation of progressive disease or death, whichever occurs first.
Progression-Free Survival (PFS) as assessed by an IRC according to the 2014 International Working Group (IWG) Lugano Criteria (Cheson, 2014). | Start of treatment up to 21 months
  PFS per IRC. PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the IRC or death from any cause, whichever occurs first.
Complete Response (CR) Rate as assessed by an IRC according to the 2014 International Working Group (IWG) Lugano Criteria (Cheson, 2014). | Start of treatment to 21 months
  CR rate per IRC according to the 2014 IWG Lugano criteria (Cheson, 2014)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Northwestern University, Evanston, Illinois
  - Henry Ford Health, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas, M. D. Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas